CLINICAL TRIAL: NCT06601309
Title: Biomarker Based Neoadjuvant Strategies for Locally Advanced Resectable Esophageal Squamous Cell Carcinoma: an Exploratory Phase II Single-arm Clinical Study
Brief Title: Biomarker Based Neoadjuvant Strategies for Locally Advanced Resectable ESCC
Acronym: ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Yong Yang, Principal Investigator, Fujian Medical University Union Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIONS-R
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Cancer; Neoadjuvant Therapy; Pathological Complete Response (pCR); Immunotherapy; Chemoradiotherapy; Biomarkers
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — TP protocol; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Intervention Model Description: This parallel assignment interventional study evaluates the efficacy and safety of biomarker-based neoadjuvant treatments in resectable locally advanced esophageal squamous cell carcinoma (ESCC). Patients are stratified by PD-L1 expression (CPS) into three groups:
  1. High PD-L1 Expression (CPS ≥ 20) Neoadjuvant immunotherapy alone.
  2. Moderate PD-L1 Expression (CPS 10-20): Neoadjuvant chemotherapy combined with immunotherapy.
  3. Low PD-L1 Expression (CPS < 10): Standard neoadjuvant chemoradiotherapy.
  All treatments are followed by surgical resection. The primary endpoint is the pathological complete response (pCR) rate post-surgery. Secondary endpoints include treatment-related toxicity, R0 resection rate, and 3-year disease-free survival (DFS). Exploratory endpoints include identifying molecular biomarkers linked to treatment efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High PD-L1 Expression Group (CPS ≥ 20) (Experimental): Patients with high PD-L1 expression (CPS ≥ 20) will receive neoadjuvant immunotherapy alone. This treatment consists of serplulimab for 2 cycles.
  Interventions: Drug: Serplulimab
- Moderate PD-L1 Expression Group (CPS 10-20) (Experimental): Patients with moderate PD-L1 expression (CPS 10-20) will receive neoadjuvant chemotherapy combined with immunotherapy. This includes paclitaxel and cisplatin along with serplulimab for 2 cycles.
  Interventions: Drug: Serplulimab; Drug: Paclitaxel+Cisplatin (Neoadjuvant Chemotherapy)
- Low PD-L1 Expression Group (CPS < 10) (Experimental): Patients with low PD-L1 expression (CPS < 10) will receive standard neoadjuvant chemoradiotherapy. This includes paclitaxel and cisplatin along with radiotherapy (40 Gy in 20 fractions over 4 weeks).
  Interventions: Drug: Paclitaxel+Cisplatin(Concurrent Chemoradiotherapy); Radiation: Radiotherapy

INTERVENTIONS:
Drug: Serplulimab — Serplulimab (300 mg) administered intravenously on day 1 of each 21-day cycle for 2 cycles.
  Arms: High PD-L1 Expression Group (CPS ≥ 20); Moderate PD-L1 Expression Group (CPS 10-20)
Drug: Paclitaxel+Cisplatin (Neoadjuvant Chemotherapy) — Paclitaxel (175 mg/m²) and Cisplatin (75 mg/m²) administered intravenously on day 1 of each 21-day cycle for 2 cycles as part of neoadjuvant chemotherapy.
  Arms: Moderate PD-L1 Expression Group (CPS 10-20)
Drug: Paclitaxel+Cisplatin(Concurrent Chemoradiotherapy) — Paclitaxel (50 mg/m²) and Cisplatin (25 mg/m²) administered intravenously on days 1, 8, 15, and 22 of a 4-week cycle as part of concurrent chemoradiotherapy.
  Arms: Low PD-L1 Expression Group (CPS < 10)
Radiation: Radiotherapy — Radiotherapy at a dose of 40 Gy, delivered in 20 fractions over 4 weeks.
  Arms: Low PD-L1 Expression Group (CPS < 10)

SUMMARY:
This study aims to evaluate the impact of the neoadjuvant treatment strategy based on CPS score on the pathological complete response (pCR) rate in patients with resectable locally advanced esophageal cancer.

DETAILED DESCRIPTION:
Esophageal cancer is a malignant tumor with a high incidence in China, with most patients diagnosed at the advanced stage. Traditional treatment modalities include surgery, chemoradiotherapy, and chemotherapy. However, under current standard treatments, approximately 50% of patients remain incurable, primarily due to postoperative recurrence and distant metastasis. Therefore, seeking a new treatment strategy to improve efficacy is crucial.

This clinical trial aims to evaluate the use of immune checkpoint inhibitors in neoadjuvant therapy based on CPS scoring to enhance the pathologic complete response (pCR) rate. Patients pathologically confirmed with esophageal squamous cell carcinoma (ESCC) will undergo surgical assessment for operability. Eligible patients will further undergo CPS testing and will receive different neoadjuvant treatment strategies based on CPS results: patients with CPS ≥20 will receive neoadjuvant immunotherapy alone; CPS 10-20 patients will receive neoadjuvant chemotherapy followed by immunotherapy; and CPS <10 patients will receive standard neoadjuvant chemoradiotherapy.

After completing neoadjuvant therapy, patients will rest for 4-6 weeks before undergoing curative surgery, which will be reassessed by thoracic surgeons for R0 resection feasibility preoperatively. Postoperatively, pathological evaluation will assess the pCR rate and other secondary study endpoints, with the most severe toxicities included in the analysis.

This study anticipates a group-wide pCR rate of 45% based on a PD-L1 biomarker-guided neoadjuvant treatment strategy. The trial is designed to exclude a pCR rate of 30% or lower using a one-sided 95% confidence interval (α set at 0.025) and 80% statistical power, with a total sample size of 90. The null hypothesis will be rejected if fewer than 34 patients achieve pCR in the entire cohort.

Based on reference studies (EC-CRT-001, ESCORT-1, JUPITER-06, and KEYNOTE-590) and CPS distribution data for esophageal squamous cell carcinoma from our institution, it is expected that the proportions of patients with CPS ≥20, 10-20, and <10 will be 10%, 40%, and 50%, respectively, corresponding to 9, 36, and 45 eligible patients for each group. It is anticipated that biological specimens will be obtained from more than 30 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Histologically confirmed esophageal squamous cell carcinoma (ESCC).
2. Stage: Resectable locally advanced ESCC (clinical stage II-III according to the AJCC/UICC 8th edition).
3. Age: 18-75 years old.
4. Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
5. PD-L1 Expression: Available PD-L1 expression level (CPS).
6. Surgical Eligibility: Assessed as eligible for surgical resection by a thoracic surgeon.
7. Laboratory Requirements:

   * Adequate bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, Platelets ≥ 100 x 10^9/L, Hemoglobin ≥ 9 g/dL.
   * Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), AST and ALT ≤ 2.5 x ULN.
   * Adequate renal function: Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 60 mL/min.
8. Informed Consent: Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Distant Metastasis: Presence of distant metastasis.
2. Other Malignancies: History of other malignancies within the past 5 years, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin carcinoma, or other localized non-invasive malignancy.
3. Autoimmune Diseases: History of active autoimmune diseases requiring systemic treatment within the past 2 years.
4. Infections: Active infection requiring systemic therapy.
5. Uncontrolled Conditions: Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Previous Treatment: Previous treatment with anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies.
7. Pregnancy and Lactation: Pregnant or breastfeeding women. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization.
8. Allergies: Known allergy or hypersensitivity to study drugs or any excipient of these medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | after the pathological examination of surgical speciments within 14 days after the operation
  The proportion of patients achieving a pathological complete response (pCR) after neoadjuvant treatment and surgical resection. pCR is defined as the absence of any residual invasive cancer in the resected esophagus and all sampled lymph nodes (ypT0N0) based on hematoxylin and eosin staining.

SECONDARY OUTCOMES:
R0 Resection Rate | after the pathological examination of surgical speciments ie within 14 days after the operation
  The proportion of patients achieving an R0 resection, defined as a microscopically margin-negative resection with no residual tumor at the resection margins.
Treatment-Related Toxicity | From the start of treatment to 30 days post-surgery
  The incidence and severity of treatment-related adverse events, graded according to CTCAE 5.0. This includes adverse events related to Serplulimab, Paclitaxel, Cisplatin, and radiotherapy, as well as surgical complications.
3-Year Disease-Free Survival (DFS) | 36 months after treatment completion
  The percentage of patients who remain disease-free three years after surgical resection. DFS is defined as the time from R0 resection to the first occurrence of disease recurrence or death from any cause.
Tumor Mutational Burden (TMB) | 36 months after treatment completion.
  Tumor mutational burden (TMB) score as measured in tumor tissue samples.
Microsatellite Instability (MSI) | 36 months after treatment completion
  Percentage of patients with high microsatellite instability (MSI-H) in tumor tissue
Circulating Tumor DNA (ctDNA) | 36 months after treatment completion
  Change in circulating tumor DNA (ctDNA) levels as measured by liquid biopsy.
major pathological response | Patients were evaluated 2 to 4 weeks postoperatively.
  tumor regression ≥90%

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No